CLINICAL TRIAL: NCT05703789
Title: Oral Health in Patients With Severe Eating Disorders An Interview, Questionnaire and Intervention Study With a Focus on Quality of Life
Brief Title: Oral Health in Patients With Severe Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Public Dental Health Service in Stockholm AB (Unknown)
Responsible Party: Principal Investigator, Göran Dahllöf, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03601
Record Dates: First submitted 2022-11-23; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Oral Health Related Quality of Life
Keywords: prosthetic rehabilitation; eating disorder; quality of life; dental
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either oral rehabilitation or a waiting-list condition for 4-6 months. Patients receiving dental treatment will be allocated to one of two different treatment groups based on individual treatment need and proven experience. Patients in group 1 will be treated with minimal invasive treatment, with restorative composite fillings. Patients in group 2 will be treated with prosthetic rehabilitation, dental crowns. Patients that are randomized to no dental treatment will act as controls. The overall treatment results will be followed up after 4, 12 and 24 months. After the 4-6-month follow-up, the corresponding control patient from the waiting list will receive requisite dental treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral rehabilitation (Experimental): Name Oral rehabilitation. Patients receiving dental treatment will be allocated to one of two different treatment groups based on individual treatment need and proven experience. Patients in group 1 will be treated with minimal invasive treatment, with restorative composite fillings. Patients in group 2 will be treated with prosthetic rehabilitation, dental crowns.
  Interventions: Procedure: Dental rehabilitation with either composite resin of crown therapy
- Waiting list (Other): Name: Waiting list. Patients in waiting list will receive no treatment. After four months they will be offered to be included in the oral rehabilitation arm.
  Interventions: Other: Waiting list

INTERVENTIONS:
Procedure: Dental rehabilitation with either composite resin of crown therapy — Patients in group 1 will be treated with minimal invasive treatment, with restorative composite fillings. Patients in group 2 will be treated with prosthetic rehabilitation, dental crowns.
  Arms: Oral rehabilitation
Other: Waiting list — Waiting list. Patients randomized to this group will not receive any intervention but answer questionnaires after 4 months on waiting list
  Arms: Waiting list

SUMMARY:
The overall aim of the research project is to assess whether the quality of life of patients with severe eating disorders is improved by dental treatment.

Patients diagnosed with anorexia nervosa, bulimia nervosa or non-specific binge eating disorder with extensive dental treatment need will be treated with resin composite restorations or prosthetic therapy. The primary outcome measures is oral health related quality of life. Secondary are orofacial functions and oral esthetics. Patients will be compared to a waiting list.

DETAILED DESCRIPTION:
III. Do patients with severe eating disorders experience a difference in quality of life following oral rehabilitation with minimal invasive treatment or prosthetic treatment? - A prospective clinical 2-year follow-up

HYPOTHESIS The hypothesis is that patients with severe eating disorders do not exhibit any difference in terms of Oral Health Related Quality of Life following oral rehabilitation or not (null hypotheses).

PATIENTS

Patients diagnosed with anorexia nervosa, bulimia nervosa or non-specific binge eating disorder who meet the inclusion criteria will consecutively be offered to participate in the study during years 2022-2023. Spoken and written information will be given, and written consent will be obtained from all participants prior to study start.

STUDY DESIGN We will conduct a randomized controlled clinical study that examines the effect of two dental treatments on Oral Health Related Quality of Life (OHRQoL) in patients with severe anorexia nervosa, bulimia nervosa or non-specific binge eating disorder. 90 patients will be randomized 2:1 to treatment or no treatment.

Inclusion criteria Patients diagnosed with anorexia nervosa, bulimia nervosa or non-specific binge eating disorder for a minimum of 10 years = definition of a "severe" eating disorder where extensive dental damage can be anticipated to find.

Need of dental treatment of at least six teeth in one jaw, since dental treatment need of ≤ than six teeth per jaw is not expected to cause a noticeable change in OHRQoL.

Exclusion criteria Age <18 years or patients unable to provide informed consent.

EXPOSURE/INTERVENTION Patients will be randomized to either oral rehabilitation or a waiting-list condition for 4-6 months. Patients receiving dental treatment will be allocated to one of two different treatment groups based on individual treatment need and proven experience. Patients in group 1 will be treated with minimal invasive treatment, with restorative composite fillings. Patients in group 2 will be treated with prosthetic rehabilitation, dental crowns. Patients that are randomized to no dental treatment will act as controls. The overall treatment results will be followed up after 4, 12 and 24 months. After the 4-6-month follow-up, the corresponding control patient from the waiting list will receive requisite dental treatment.

Adverse events Data of adverse events will be recorded post-dental treatment using an online questionnaire where participants will be able to describe any adverse event during treatment in detail. Patients who report at least one adverse event will receive follow-up questions about the duration and intensity of the event.

DATA COLLECTION The primary outcome, OHRQoL will be evaluated by means of a validated psychometrical instrument for reporting this: oral health impact (OHIP-49). Longitudinal comparison in patients receiving no treatment (controls). and treatment OHIP-49 is a survey with 49 questions divided into 7 subgroups: Functional limitation, Physical pain, Psychologic disability, Social disability, Handicap, Orofacial Appearance and Psychosocial Impact. The categories will be graded from 0 to 4 on a Likert Scale (never = 0, seldom= 1, sometimes = 2, fairly often = 3, and very often = 4). The internal reliability, and test/retest reliability and validity of the OHIP-49 has previously been established. Since OHIP-49 measures capture both improvements and declines in oral health status, the instrument enables the possibility to conceptualize and analyze change longitudinally. Additional outcome measures are orofacial function (JFL-S) and oral aesthetics (OES).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with anorexia nervosa, bulimia nervosa or non-specific binge eating disorder for a minimum of 10 years = definition of a "severe" eating disorder where extensive dental damage can be anticipated to find.
* Need of dental treatment of at least six teeth in one jaw,

Exclusion Criteria:

* Age <18 years or patients unable to provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life OHIP-49 | Before treatment
  OHIP-49 is a survey with 49 questions divided into 7 subgroups: Functional limitation, Physical pain, Psychologic disability, Social disability, Handicap, Orofacial Appearance and Psychosocial Impact. The categories will be graded from 0 to 4 on a Likert Scale (never = 0, seldom= 1, sometimes = 2, fairly often = 3, and very often = 4). The internal reliability, and test/retest reliability and validity of the OHIP-49 has previously been established. Since OHIP-49 measures capture both improvements and declines in oral health status, the instrument enables the possibility to conceptualize and analyze change longitudinally.
Oral health related quality of life OHIP-49 | 4 months
  OHIP-49 is a survey with 49 questions divided into 7 subgroups: Functional limitation, Physical pain, Psychologic disability, Social disability, Handicap, Orofacial Appearance and Psychosocial Impact. The categories will be graded from 0 to 4 on a Likert Scale (never = 0, seldom= 1, sometimes = 2, fairly often = 3, and very often = 4). The internal reliability, and test/retest reliability and validity of the OHIP-49 has previously been established. Since OHIP-49 measures capture both improvements and declines in oral health status, the instrument enables the possibility to conceptualize and analyze change longitudinally.
Oral health related quality of life OHIP-49 | 12 months
  OHIP-49 is a survey with 49 questions divided into 7 subgroups: Functional limitation, Physical pain, Psychologic disability, Social disability, Handicap, Orofacial Appearance and Psychosocial Impact. The categories will be graded from 0 to 4 on a Likert Scale (never = 0, seldom= 1, sometimes = 2, fairly often = 3, and very often = 4). The internal reliability, and test/retest reliability and validity of the OHIP-49 has previously been established. Since OHIP-49 measures capture both improvements and declines in oral health status, the instrument enables the possibility to conceptualize and analyze change longitudinally.
Oral health related quality of life OHIP-49 | 24 months
  OHIP-49 is a survey with 49 questions divided into 7 subgroups: Functional limitation, Physical pain, Psychologic disability, Social disability, Handicap, Orofacial Appearance and Psychosocial Impact. The categories will be graded from 0 to 4 on a Likert Scale (never = 0, seldom= 1, sometimes = 2, fairly often = 3, and very often = 4). The internal reliability, and test/retest reliability and validity of the OHIP-49 has previously been established. Since OHIP-49 measures capture both improvements and declines in oral health status, the instrument enables the possibility to conceptualize and analyze change longitudinally.

SECONDARY OUTCOMES:
Orofacial function (JFL-S) | Before treatment
  JFLS is an instrument used for evaluating functional limitations. It measures mastication, vertical jaw mobility, verbal and emotional expression as well as miscellaneous functions such as swallow food and yawn. This instrument is a 20-item questionnaire which exhibits good reliability and validity and has been shown to be useful in assessing functional limitations of the jaws [18]. Subjects rate their jaw functional limitations on a numeric rating scale (0- 'no limitation', 10- 'extreme limita- tion'). Total score can range from 0 to 200, where 200 is the highest score which indicates extreme limitations.
Orofacial function (JFL-S) | 4 months
  JFLS is an instrument used for evaluating functional limitations. It measures mastication, vertical jaw mobility, verbal and emotional expression as well as miscellaneous functions such as swallow food and yawn. This instrument is a 20-item questionnaire which exhibits good reliability and validity and has been shown to be useful in assessing functional limitations of the jaws [18]. Subjects rate their jaw functional limitations on a numeric rating scale (0- 'no limitation', 10- 'extreme limita- tion'). Total score can range from 0 to 200, where 200 is the highest score which indicates extreme limitations.
Orofacial function (JFL-S) | 12 months
  JFLS is an instrument used for evaluating functional limitations. It measures mastication, vertical jaw mobility, verbal and emotional expression as well as miscellaneous functions such as swallow food and yawn. This instrument is a 20-item questionnaire which exhibits good reliability and validity and has been shown to be useful in assessing functional limitations of the jaws [18]. Subjects rate their jaw functional limitations on a numeric rating scale (0- 'no limitation', 10- 'extreme limita- tion'). Total score can range from 0 to 200, where 200 is the highest score which indicates extreme limitations.
Orofacial function (JFL-S) | 24 months
  JFLS is an instrument used for evaluating functional limitations. It measures mastication, vertical jaw mobility, verbal and emotional expression as well as miscellaneous functions such as swallow food and yawn. This instrument is a 20-item questionnaire which exhibits good reliability and validity and has been shown to be useful in assessing functional limitations of the jaws [18]. Subjects rate their jaw functional limitations on a numeric rating scale (0- 'no limitation', 10- 'extreme limita- tion'). Total score can range from 0 to 200, where 200 is the highest score which indicates extreme limitations.
Oral aesthetics (OES). | Before treatment
  OES is an instrument used to evaluate self-perceived orofacial aesthetics and the reliability and validity has been investigated previously [19,26]. The instrument is an eight- item questionnaire which measures aesthetic components such as appearance of the face, facial profile, mouth, align- ment, tooth shape, tooth colour and gum as well as a gen- eral orofacial aesthetic assessment. Subjects respond on a 0-10 numeric rating scale (0- 'very dissatisfied', 10- 'very sat- isfied') or mark the answer 'not applicable' if they do not wish to answer. The total score can range from 0 to 70, where 70 is the highest score which indicates very high satis- faction. Subjects were allowed to ask questions if needed but answered the questionnaires on their own.
Oral aesthetics (OES). | 4 months
  OES is an instrument used to evaluate self-perceived orofacial aesthetics and the reliability and validity has been investigated previously [19,26]. The instrument is an eight- item questionnaire which measures aesthetic components such as appearance of the face, facial profile, mouth, align- ment, tooth shape, tooth colour and gum as well as a gen- eral orofacial aesthetic assessment. Subjects respond on a 0-10 numeric rating scale (0- 'very dissatisfied', 10- 'very sat- isfied') or mark the answer 'not applicable' if they do not wish to answer. The total score can range from 0 to 70, where 70 is the highest score which indicates very high satis- faction. Subjects were allowed to ask questions if needed but answered the questionnaires on their own.
Oral aesthetics (OES). | 12 months
  OES is an instrument used to evaluate self-perceived orofacial aesthetics and the reliability and validity has been investigated previously [19,26]. The instrument is an eight- item questionnaire which measures aesthetic components such as appearance of the face, facial profile, mouth, align- ment, tooth shape, tooth colour and gum as well as a gen- eral orofacial aesthetic assessment. Subjects respond on a 0-10 numeric rating scale (0- 'very dissatisfied', 10- 'very sat- isfied') or mark the answer 'not applicable' if they do not wish to answer. The total score can range from 0 to 70, where 70 is the highest score which indicates very high satis- faction. Subjects were allowed to ask questions if needed but answered the questionnaires on their own.
Oral aesthetics (OES). | 24 months
  OES is an instrument used to evaluate self-perceived orofacial aesthetics and the reliability and validity has been investigated previously [19,26]. The instrument is an eight- item questionnaire which measures aesthetic components such as appearance of the face, facial profile, mouth, align- ment, tooth shape, tooth colour and gum as well as a gen- eral orofacial aesthetic assessment. Subjects respond on a 0-10 numeric rating scale (0- 'very dissatisfied', 10- 'very sat- isfied') or mark the answer 'not applicable' if they do not wish to answer. The total score can range from 0 to 70, where 70 is the highest score which indicates very high satis- faction. Subjects were allowed to ask questions if needed but answered the questionnaires on their own.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastman Dental Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Result] Larsson P, John MT, Nilner K, Bondemark L, List T. Development of an Orofacial Esthetic Scale in prosthodontic patients. Int J Prosthodont. 2010 May-Jun;23(3):249-56. PMID 20552092